CLINICAL TRIAL: NCT05902000
Title: Stent Implantation Versus Balloon Dilation for Acute Anterior Circulation Tandem Occlusion: A Multicenter, Prospective, Randomized, Open-label, Blinded End-point Trial
Brief Title: Stent Implantation Versus Balloon Dilation for Acute Anterior Circulation Tandem Occlusion
Acronym: START
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xueli Cai (Other Government)
Responsible Party: Sponsor-Investigator, Xueli Cai, Chief physician, Lishui Municipal Central Hospital
Organization: Lishui Municipal Central Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WKJ-ZJ-2327
Record Dates: First submitted 2023-04-05; First posted 2023-06-13 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Thrombectomy; Tandem Occlusion; Stroke
Keywords: tandem occlusion; anterior circulation; stent implantation; balloon dilation; randomized controlled trial
MeSH Terms: conditions — Stroke | interventions — Thrombectomy

STUDY DESIGN:
Intervention Model Description: Carotid artery stenting after intracranial or middle cerebral artery embolization and balloon dilation of the extracranial segment of the ipsilateral internal carotid artery
Who Masked: Outcomes Assessor
Masking Description: 1. Randomization results are known only to the patients themselves and the treating physicians. Baseline and in-hospital visits related to the study endpoint should be evaluated by a third party who is unknown to the patients' grouping and actual treatment status.2. Visits to the primary endpoint were conducted by trained third-party personnel. Standardized visits were conducted under the premise of unknown patient randomization and actual treatment status, and follow-up reports were prepared.3. All research-related image data will be collected for centralized interpretation. The images at each site were interpreted independently, and the readers were not aware of the patient's baseline condition, treatment received (except the images during baseline surgical treatment), and prognosis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrombectomy + Carotid Stenting (Experimental): After emergency admission,intravenous thrombolysis will be administered if possible. Standard endovascular thrombectomy (EMT) and balloon angioplasty will be performed. The method of EMT and the order of endovascular treatment were selected by each center. After EMT and balloon angioplasty, patients with eTICI≥2b_50 were maintained for more than 10 minutes for randomization. In the intervention arm, emergent carotid stenting will be performed. Standardized treatment with antiplatelet and other drugs will be given. A loading dose of antiplatelet agents (aspirin 300 mg and clopidogrel 300 mg) or Tirofiban was given as an intraoperative drug treatment to endovascular therapy prior to emergency balloon dilation or stenting. Intravenous sedation or general anesthesia will be permitted.
  Oral dual antiplatelet treatment for more than 1 month. Tirofiban is maintained for 24-48 hours, overlapping with oral antiplatelet for 4-6 hours, after excluding intracranial hemorrhage.
  Interventions: Device: Carotid Stenting; Procedure: Thrombectomy; Drug: Dual antiplatelet treatment; Drug: Intraoperative Drug Treatment
- Thrombectomy alone (No Intervention): Intracranial thrombectomy alone（balloon dilation of the ipsilateral internal carotid artery if necessary）

INTERVENTIONS:
Device: Carotid Stenting — Emergent carotid stenting will be performed if the patient is randomized in the intervention arm. The order to treat (head first or neck first) the extracranial carotid artery lesion will be left to the interventionist discretion.
  Arms: Thrombectomy + Carotid Stenting
Procedure: Thrombectomy — Intracranial thrombectomy is an endovascular procedure. In the experimental group, thrombectomy will be completed with extracranial carotid stenting.
  Arms: Thrombectomy + Carotid Stenting
Drug: Dual antiplatelet treatment — Dual antiplatelet therapy is administered after 24 hours of imaging follow-up excluding intracranial hemorrhagic complications. Aspirin Enteric-coated Tablets (Bay Aspirin) 100mg once a night+Clopidogrel Sulfate Tablets (Plavix) 75mg once daily. If there is no contraindication, maintain for more than 1 month, then adjust the dosing regimen according to the guidelines.
  Arms: Thrombectomy + Carotid Stenting
Drug: Intraoperative Drug Treatment — Tirofiban is used as an adjunct to endovascular therapy. The currently recommended dosing regimen is a combined intra-catheter arterial administration of a loading dose of 0.4 μg/(kg-min) for 30 min (total dose not to exceed 1 mg)， followed by intravenous pumping of 0.1μg/(kg-min) for 24-48h, and adjustment of dosing in conjunction with CT.
  Arms: Thrombectomy + Carotid Stenting

SUMMARY:
1. To evaluate whether stent implantation on the ipsilateral extracranial segment, after intracranial thrombectomy successful recanalization compared with balloon angioplasty (eTICI≥2b_50) for acute anterior circulation tandem lesions within 24h of onset, can improve neurological functional outcomes(mRS≤2).
2. To evaluate whether stent implantation on the ipsilateral extracranial segment, after intracranial thrombectomy successful recanalization compared with balloon angioplasty (eTICI≥2b_50) for acute anterior circulation tandem lesions within 24h of onset, can increase the risk of symptomatic intracranial hemorrhage.

DETAILED DESCRIPTION:
The study was a prospective, randomized, open-label, blinded end-point Clinical Trial.

Subjects were randomized 1:1 according to inclusion and exclusion criteria into a trial group (acute phase extracranial vascular stent implantation group) and a control group (acute phase non-extracranial vascular stent implantation group). Randomization was performed for 90d and 180d for the follow-up to collect primary and secondary efficacy and safety indicators.

ELIGIBILITY:
General inclusion criteria

1. Age 18-85 years old;
2. Acute ischemic stroke and the onset time within 24h;
3. Pre-stroke mRS 0-1;
4. NIHSS score of 6-30 before randomization;
5. Completed randomization within 24h after stroke onset；
6. Subjects are able to sign an informed consent in person or by the legal representative

Imaging Inclusion Criteria:

1. Satisfy one of the following criteria:①Within 6 hours of onset, imaging confirmed occlusion of the acute anterior circulation internal carotid artery or the M1 / M2 segment of the middle cerebral artery；②Within 6-16 hours of onset, imaging confirmed acute occlusion of anterior circulation internal carotid artery or M1 / M2 segment of middle cerebral artery followed by DAWN or DEFUSE-3 criteria；③In patients with 16 to 24 hours of onset, imaging confirmed intracranial occlusion of the acute anterior circulation internal carotid artery or M1 / M2 segment of the middle cerebral artery followed by DAWN criteria.
2. Extracranial segment stenosis ≥70% or occlusion in tandem lesions.
3. ASPECT score ≥ 6 points.
4. eTICI≥2b_50 after middle cerebral artery thrombectomy and extracranial balloon dilatation in 10min.

General Exclusion Criteria:

Participating in other clinical trials; 2.It is planned to carry out selective internal carotid artery stent implantation within 3 months; 3.Intracranial hemorrhage, subarachnoid hemorrhage within 3 months; previous brain tumor (with space-occupying effect).

4.Parenchymal organ surgery or biopsy were performed last 1 month; Any active or recent bleeding (gastrointestinal, urinary, etc.); Parenchymal organ surgery and biopsy were performed last 1 month 5.Difficult to control hypertension: systolic blood pressure> 185mmHg and/ or diastolic blood pressure> 110mmHg.

6.Severe active bleeding or known significant bleeding tendency: platelet count <100X109/L; heparin within 48 hours before surgery, and APTT≥35s; oral warfarin, and INR> 1.7; direct thrombin or factor Xa inhibitors, such as apixaban tablets, rivaroxaban tablets and dabigatran (patients with no history of abnormal coagulation or suspected abnormal coagulation function do not need laboratory results of INR or APTT before enrollment）.

7.Severe heart, liver, kidney, and other organ insufficiencies (glomerular filtration rate <30 ml/min or blood creatinine> 220μmol/L(2.5mg/dl)).

8.Patients occurred acute ischemic cerebral infarction within 48 hours after percutaneous coronary or cerebrovascular intervention or major surgery (if more than 48h, patients may be enrolled).

9. The patient has a history of cerebral vasculitis with clear evidence; 10. Patients with pre-onset neurological or psychiatric disorders that affect the assessment of their condition 11.Women who are known to be pregnant or lactating. 12.Known severe allergy to contrast agents (except for mild rash allergy) 13.Expected survival time less than 1 year (such as combined malignancy, severe cardiopulmonary disease, etc.) 14.Patients unable to complete the follow up (e. g., no fixed residence, overseas patients, etc.).

Imaging exclusion criterias:

1. Imaging confirmed the posterior circulatory lesions.
2. Midline displacement of the brain or brain herniation, ventricular occupancy
3. New onset bilateral acute stroke or multiple intracranial macrovascular occlusions.
4. Patients with vascular variants that are difficult to treat with endovascular therapy as displayed by CTA/MRA;
5. The ipsilateral middle cerebral artery and anterior cerebral occlusion were combined.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of functional independence | at 90±7 days
  Rate of functional independence defined as a modified Rankin Scale (mRS) score 0-2 at 90 (±7 days) (blind and independent evaluation) The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire. The Modified Rankin Score (mRS) is the most widely used outcome measure in stroke clinical trials. Standardized interviews to obtain a mRS score are recommended at 3 months (90 days) following hospital discharge.
Rate of symptomatic intracranial hemorrhage | at 36 hours (±12 hours)
  Rate of symptomatic intracerebral hemorrhage at CT (Computerized Tomography) or MRI (Magnetic Resonance Imaging) at 36 hours (±12 hours) according to the Heidelberg classification (independent imaging core laboratory).

SECONDARY OUTCOMES:
The expanded treatment in cerebral infarction (eTICI) score | at the end of the endovascular procedure
  eTICI score (0,1,2a,2a_50,2a_67,2c,3) : Grade 0 : no perfusion Grade 1: penetration with minimal perfusion Grade 2a: partial filling of 1-49% of the vascular territory Grade 2b_50 : partial filling of 50-66% of the vascular territory Grade 2b_67: partial filling of 67-89% of the vascular territory Grade 2c: partial filling of 90-99% of the vascular territory Grade 3 : complete perfusion
Ipsilateral carotid residual stenosis rate | at the end of the endovascular procedure
  The extracranial stenosis was assessed by using criteria from the North American Symptomatic Carotid Endarterectomy Trial (NASCET). The residual stenosis rate of the ipsilateral internal carotid artery was assessed according to the last DSA angiography of the procedure.
The National Institutes of Health Stroke Scale (NIHSS) score | at 36 hours (±12 hours)
  National Institutes of Health Stroke Scale (NIHSS) score. The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The single patient assessment requires less than 10 minutes to complete. The evaluation of stroke severity depends upon the ability of the observer to accurately and consistently assess the patient.
  Higher scores mean a worse outcome.
Proportion of NIHSS scores 0-1 | at 36 hours (±12 hours)
  The proportion of patients with an NIHSS score of 0-1
  National Institutes of Health Stroke Scale (NIHSS) score. The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The single patient assessment requires less than 10 minutes to complete. The evaluation of stroke severity depends upon the ability of the observer to accurately and consistently assess the patient.
  Higher scores mean a worse outcome.
Change in National Institutes of Health Stroke Scale (NIHSS) score | at 36 hours (±12 hours)
  The proportion of patients with an NIHSS score reduction of ≥4 points after randomization compared to baseline.
  NIHSS is 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss.
  A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items.
  Higher scores mean a worse outcome.
Rate of carotid stenosis | at 5-7days or discharge
  The extracranial stenosis was assessed by using criteria from the North American Symptomatic Carotid Endarterectomy Trial (NASCET) confirmed by cervical vascular ultrasound.
The NIHSS score | at 5-7days or discharge
  The NIHSS score
  NIHSS is 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss.
  A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items.
  Higher scores mean a worse outcome.
The mRS scores | at 90±7days and 180±14 days
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire. The Modified Rankin Score (mRS) is the most widely used outcome measure in stroke clinical trials. Standardized interviews to obtain a mRS score are recommended at 3 months (90 days) following hospital discharge.
Proportion of mRS score 0-3 | at 90±7days and 180±14 days
  The Modified Rankin Score (mRS) is a 6-point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire. The Modified Rankin Score (mRS) is the most widely used outcome measure in stroke clinical trials. Standardized interviews to obtain an mRS score are recommended at 3 months (90 days) following hospital discharge.
  Higher scores mean a worse outcome.
All-cause mortality | at 90±7days
  Rate of mortality at 90±14 days.
Rate of asymptomatic intracranial hemorrhage | at 36 hours (±12 hours)
  Rate of symptomatic intracerebral hemorrhage at CT (Computerized Tomography) or MRI (Magnetic Resonance Imaging) at 36 hours (±12 hours) according to the Heidelberg classification (independent imaging core laboratory).
The incidence of adverse events. | at 90±7days and 180±14 days
  Any adverse medical event, whether causally related to the trial or not, that occurred between the start of patient randomization and the last follow-up visit was judged as an adverse event. The incidence of non-hemorrhagic adverse events.
The incidence of serious adverse events. | at 90±7days and 180±14 days
  A serious adverse event is defined as an adverse event that results in
  1. Resulting in death;
  2. Life-threatening (means that the subject is at risk of death at the time of an adverse event. It does not refer to those adverse events that could lead to death if the condition were assumed to be worse);
  3. Requires hospitalization or prolonged hospitalization;
  4. Resulting in persistent or severe disability or dysfunction
  5. Resulting in a congenital anomaly or birth defect;
  6. Medical events that, in the opinion of the investigator, can be judged as serious adverse events.
  The incidence of non-hemorrhagic serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Li X Cai, Principal Investigator — Lishui Municipal Hospital
Locations (1):
- Lishui Municipal Hospital, Lishui, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berkhemer OA, Majoie CB, Dippel DW; MR CLEAN Investigators. Endovascular therapy for ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2363. doi: 10.1056/NEJMc1504715. No abstract available. PMID 26061844
- [Result] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Result] Campbell BC, Mitchell PJ, Kleinig TJ, Dewey HM, Churilov L, Yassi N, Yan B, Dowling RJ, Parsons MW, Oxley TJ, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Priglinger M, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke with perfusion-imaging selection. N Engl J Med. 2015 Mar 12;372(11):1009-18. doi: 10.1056/NEJMoa1414792. Epub 2015 Feb 11. PMID 25671797
- [Result] Saver JL, Goyal M, Bonafe A, Diener HC, Levy EI, Pereira VM, Albers GW, Cognard C, Cohen DJ, Hacke W, Jansen O, Jovin TG, Mattle HP, Nogueira RG, Siddiqui AH, Yavagal DR, Baxter BW, Devlin TG, Lopes DK, Reddy VK, du Mesnil de Rochemont R, Singer OC, Jahan R; SWIFT PRIME Investigators. Stent-retriever thrombectomy after intravenous t-PA vs. t-PA alone in stroke. N Engl J Med. 2015 Jun 11;372(24):2285-95. doi: 10.1056/NEJMoa1415061. Epub 2015 Apr 17. PMID 25882376
- [Result] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Result] Nogueira RG, Jadhav AP, Haussen DC, Bonafe A, Budzik RF, Bhuva P, Yavagal DR, Ribo M, Cognard C, Hanel RA, Sila CA, Hassan AE, Millan M, Levy EI, Mitchell P, Chen M, English JD, Shah QA, Silver FL, Pereira VM, Mehta BP, Baxter BW, Abraham MG, Cardona P, Veznedaroglu E, Hellinger FR, Feng L, Kirmani JF, Lopes DK, Jankowitz BT, Frankel MR, Costalat V, Vora NA, Yoo AJ, Malik AM, Furlan AJ, Rubiera M, Aghaebrahim A, Olivot JM, Tekle WG, Shields R, Graves T, Lewis RJ, Smith WS, Liebeskind DS, Saver JL, Jovin TG; DAWN Trial Investigators. Thrombectomy 6 to 24 Hours after Stroke with a Mismatch between Deficit and Infarct. N Engl J Med. 2018 Jan 4;378(1):11-21. doi: 10.1056/NEJMoa1706442. Epub 2017 Nov 11. PMID 29129157
- [Result] Albers GW, Marks MP, Kemp S, Christensen S, Tsai JP, Ortega-Gutierrez S, McTaggart RA, Torbey MT, Kim-Tenser M, Leslie-Mazwi T, Sarraj A, Kasner SE, Ansari SA, Yeatts SD, Hamilton S, Mlynash M, Heit JJ, Zaharchuk G, Kim S, Carrozzella J, Palesch YY, Demchuk AM, Bammer R, Lavori PW, Broderick JP, Lansberg MG; DEFUSE 3 Investigators. Thrombectomy for Stroke at 6 to 16 Hours with Selection by Perfusion Imaging. N Engl J Med. 2018 Feb 22;378(8):708-718. doi: 10.1056/NEJMoa1713973. Epub 2018 Jan 24. PMID 29364767
- [Result] Kim YS, Garami Z, Mikulik R, Molina CA, Alexandrov AV; CLOTBUST Collaborators. Early recanalization rates and clinical outcomes in patients with tandem internal carotid artery/middle cerebral artery occlusion and isolated middle cerebral artery occlusion. Stroke. 2005 Apr;36(4):869-71. doi: 10.1161/01.STR.0000160007.57787.4c. Epub 2005 Mar 3. PMID 15746449
- [Result] Mueller-Kronast NH, Zaidat OO, Froehler MT, Jahan R, Aziz-Sultan MA, Klucznik RP, Saver JL, Hellinger FR Jr, Yavagal DR, Yao TL, Liebeskind DS, Jadhav AP, Gupta R, Hassan AE, Martin CO, Bozorgchami H, Kaushal R, Nogueira RG, Gandhi RH, Peterson EC, Dashti SR, Given CA 2nd, Mehta BP, Deshmukh V, Starkman S, Linfante I, McPherson SH, Kvamme P, Grobelny TJ, Hussain MS, Thacker I, Vora N, Chen PR, Monteith SJ, Ecker RD, Schirmer CM, Sauvageau E, Abou-Chebl A, Derdeyn CP, Maidan L, Badruddin A, Siddiqui AH, Dumont TM, Alhajeri A, Taqi MA, Asi K, Carpenter J, Boulos A, Jindal G, Puri AS, Chitale R, Deshaies EM, Robinson DH, Kallmes DF, Baxter BW, Jumaa MA, Sunenshine P, Majjhoo A, English JD, Suzuki S, Fessler RD, Delgado Almandoz JE, Martin JC, Haussen DC; STRATIS Investigators. Systematic Evaluation of Patients Treated With Neurothrombectomy Devices for Acute Ischemic Stroke: Primary Results of the STRATIS Registry. Stroke. 2017 Oct;48(10):2760-2768. doi: 10.1161/STROKEAHA.117.016456. Epub 2017 Aug 22. PMID 28830971
- [Result] Li W, Chen Z, Dai Z, Liu R, Yin Q, Wang H, Hao Y, Han Y, Qiu Z, Xiong Y, Sun W, Zi W, Xu G, Liu X. Management of acute tandem occlusions: Stent-retriever thrombectomy with emergency stenting or angioplasty. J Int Med Res. 2018 Jul;46(7):2578-2586. doi: 10.1177/0300060518765310. Epub 2018 May 4. PMID 29726291
- [Result] Feil K, Herzberg M, Dorn F, Tiedt S, Kupper C, Thunstedt DC, Papanagiotou P, Meyer L, Kastrup A, Dimitriadis K, Liebig T, Dieterich M, Kellert L; GSR investigatorsdagger. Tandem Lesions in Anterior Circulation Stroke: Analysis of the German Stroke Registry-Endovascular Treatment. Stroke. 2021 Apr;52(4):1265-1275. doi: 10.1161/STROKEAHA.120.031797. Epub 2021 Feb 16. PMID 33588589
- [Result] Zhu F, Bracard S, Anxionnat R, Derelle AL, Tonnelet R, Liao L, Mione G, Humbertjean L, Lacour JC, Hossu G, Anadani M, Richard S, Gory B. Impact of Emergent Cervical Carotid Stenting in Tandem Occlusion Strokes Treated by Thrombectomy: A Review of the TITAN Collaboration. Front Neurol. 2019 Mar 11;10:206. doi: 10.3389/fneur.2019.00206. eCollection 2019. PMID 30915023
- [Result] Pires Coelho A, Lobo M, Gouveia R, Silveira D, Campos J, Augusto R, Coelho N, Canedo A. Overview of evidence on emergency carotid stenting in patients with acute ischemic stroke due to tandem occlusions: a systematic review and meta-analysis. J Cardiovasc Surg (Torino). 2019 Dec;60(6):693-702. doi: 10.23736/S0021-9509.18.10312-0. Epub 2018 Jan 23. PMID 29363895
- [Result] Anadani M, Spiotta AM, Alawieh A, Turjman F, Piotin M, Haussen DC, Nogueira RG, Papanagiotou P, Siddiqui AH, Lapergue B, Dorn F, Cognard C, Ribo M, Psychogios MN, Labeyrie MA, Mazighi M, Biondi A, Anxionnat R, Bracard S, Richard S, Gory B; TITAN (Thrombectomy In TANdem Lesions) Investigators. Emergent Carotid Stenting Plus Thrombectomy After Thrombolysis in Tandem Strokes: Analysis of the TITAN Registry. Stroke. 2019 Aug;50(8):2250-2252. doi: 10.1161/STROKEAHA.118.024733. Epub 2019 Jun 17. PMID 31577899
- [Result] Fox AJ. How to measure carotid stenosis. Radiology. 1993 Feb;186(2):316-8. doi: 10.1148/radiology.186.2.8421726. No abstract available.